CLINICAL TRIAL: NCT02898922
Title: Robust Antibody and Cytokine Response to Hepatitis B Vaccine Among Not-in-treatment Patients With Chronic Hepatitis C：An Open-label Control Study in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong Province Centers for Disease Control and Prevention (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government); National Institutes for Food and Drug Control, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCV-001
Record Dates: First submitted 2016-09-03; First posted 2016-09-13 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Hepatitis B Vaccines
MeSH Terms: conditions — Hepatitis B

ARMS (2):
- HCV group (Experimental): Three doses of hepatitis B vaccine made by Recombinant DNA Techniques in Saccharomyces Cerevisiae (20 μg HBsAg/1.0ml per dose, Shenzhen Kangtai Biological Products Co., Ltd., Shenzhen, Guangdong Province, China) were given intramuscularly in the deltoid region to all participants at 0, 1 and 6 months respectively.
  Interventions: Biological: hepatitis B vaccine made by Recombinant DNA Techniques in Saccharomyces Cerevisiae
- Healthy control group (Active Comparator): Three doses of hepatitis B vaccine made by Recombinant DNA Techniques in Saccharomyces Cerevisiae (20 μg HBsAg/1.0ml per dose, Shenzhen Kangtai Biological Products Co., Ltd., Shenzhen, Guangdong Province, China) were given intramuscularly in the deltoid region to all participants at 0, 1 and 6 months respectively.
  Interventions: Biological: hepatitis B vaccine made by Recombinant DNA Techniques in Saccharomyces Cerevisiae

INTERVENTIONS:
Biological: hepatitis B vaccine made by Recombinant DNA Techniques in Saccharomyces Cerevisiae — 20 μg HBsAg/1.0ml per dose, Shenzhen Kangtai Biological Products Co., Ltd., Shenzhen, Guangdong Province, China

SUMMARY:
Background Hepatitis B virus (HBV) co-infection in individuals with hepatitis C virus (HCV) can enhance the severity of hepatitis and the risks of liver cirrhosis and hepatocellular carcinoma (HCC). Hepatitis B vaccine is an effective measure to prevent HBV infection. Whether patients with HCV infection have non-protective antibody responses to hepatitis B vaccination more frequently than healthy subjects is still controversial and studies about cytokine response have been seldom reported.

Methods Not-in-treatment patients with chronic HCV infection and 1:2 community/gender matched healthy control were obtained from a community-based screening. All participants received three doses of hepatitis B vaccine (20 μg HBsAg/ml/dose) on 0, 1 and 6 months schedule. Anti-HBs was tested 1 month after the third dose of vaccination and was compared between two groups. Spot-forming cells (SFCs) of interferon-γ (IFN-γ), interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-5 (IL-5) and interleukin-6 (IL-6) produced by lymphocyte were tested by enzyme-linked immunospot (ELISPOT) and were compared between two groups.

DETAILED DESCRIPTION:
Study design and participants The study was conducted in three counties (Yucheng, Xintai and Dongchangfu) of Shandong province, China, which had the highest reported HCV case numbers in the province. Potential patients with chronic HCV infection were recruited by checking the medical records of the hospitals or by inquiring of village doctors. Healthy individuals were randomly selected by 3 to 5 times of potential patients with HCV infection in the same county. Questionnaire investigation was made and blood samples were collected for each potential patient and healthy individual in the same way.

Questionnaire survey We performed a questionnaire-based survey to collect the base line information of the participants, including demographic information (age, sex, height and weight), medical history (allergy, diagnosis and treatment of chronic hepatitis C, vaccination, fever, and other acute diseases), and behavioral status (smoking, drinking, pregnancy and lactation).

Hepatitis B vaccination and follow-up Three doses of hepatitis B vaccine made by Recombinant DNA Techniques in Saccharomyces Cerevisiae (20 μg HBsAg/1.0ml per dose, Shenzhen Kangtai Biological Products Co., Ltd., Shenzhen, Guangdong Province, China) were given intramuscularly in the deltoid region to all participants at 0, 1 and 6 months respectively. Blood samples from the participants were collected one month after the first and the third dose of vaccination.

Laboratory assays and physical examination Screening test and physical examination HBsAg, anti-HBs, HBeAg, anti-HBe, anti-HBc, anti-HCV and HCV RNA were assayed for all subjects at inclusion visits; serum bilirubin, serum albumin, prothrombin time, plasma ALT and aspartate aminotransferase (AST) were detected for HCV group. HBsAg, anti-HBs, HBeAg, anti-HBe and anti-HBc were assayed by Abbott Chemiluminesent Microparticle ImmunoAssay (CMIA) (Abbott Ireland Diagnostics Division, Sligo, Ireland). Anti-HCV was measured by ELISA with a commercial kit (Intec products, INC, Xiamen, China). HCV RNA was measured by Quantitative Real-time PCR with commercially available kits (QIAGEN, Shenzhen, China). Serum bilirubin, albumin, prothrombin time, plasma ALT and AST were measured using standard reagent and methods. In order to assess disease activity, each patient with HCV infection received clinical examination, including interrogation, physical examination and ultrasonography.

Anti-HBs assay after vaccination Anti-HBs was detected using CMIA (Abbott Ireland Diagnostics Division, Sligo, Ireland) one month after the first and the third dose of vaccination. Although without serological HBV markers, subjects were defined as having a history of HBV infection or hepatitis B vaccination if anti-HBs ≥100 mIU/ml one month after the first dose of vaccination.

CMI assay Before the first dose of vaccination and one month after the third dose of vaccination, 43 subjects from HCV group and 37 subjects from healthy control group were selected randomly to isolated peripheral blood mononuclear cells (PBMCs) and tested CMI function respectively, including interferon-γ (IFN-γ), interleukin-2 (IL-2), interleukin-4 (IL-4), interleukin-5 (IL-5) and interleukin-6 (IL-6). S28-39 polypeptide, MHC class I polypeptide, MHC class II polypeptide and HBsAg were used as cell immunologic stimulant of IFN-γ respectively. Hepatitis B virus surface antigen was used as cell immunologic stimulant of IL-2, IL-4, IL-5 and IL-6. S28-39 polypeptide ，MHC class I polypeptide mixtures and MHC class II polypeptide mixtures was synthetized in BO MAI JIE Technology Co. LTD. (Beijing, China). HBsAg was supplied by Shenzhen Kangtai Biological Products Co., Ltd. (Shenzhen, China).

PBMCs separated from EDTA-anticoagulated blood were adjusted to the concentration of 2 × 106 cells /mL. 100 μL 2 × 106 cells /mL PBMCs were added in the pre-coated PVDF 96-well plates and 100 μL HBsAg S28-39 peptide (IPQSLDSWWTSL, final concentration: 10 μg/mL), 100 μL MHC class I polypeptide mixtures, 100 μL MHC class II polypeptide mixture or 100 μL HBsAg (80μg/mL) in each well. When it came to IL-2, IL-4, IL-5 and IL-6, plates were flooded with 100 μL 2 × 106 cells /mL PBMC and 100 μL HBsAg (80μg/mL) in each well. Then they were incubated at 37 °C, in a 5% CO2 and humidified incubator for 20 h (IFN-γ, IL-2) or 40 h (IL-4, IL-5 and IL-6). After incubation the plates were manipulated according to R&D ELISPOT Kit (R&D Systems, Inc.) Instruction Manual. Spot-forming Cells (SFCs) were enumerated with ImmunoSpotTM system (Cellular Technology Ltd.).

Safety assessment Participants were provided with diary cards to record the occurrence and severity of solicited local reactions at the injection site (pain, induration, erythema, edema, pruritus) during 7 days after vaccination, solicited systemic reactions (fever, headache, fatigued, cough, myalgia, asthenia, vertigo, diarrhea), and any unsolicited adverse during 29 days after vaccination.

Statistical analyses Data entry and database management were performed by EPIDATA 3.0 and Microsoft excel 2010 respectively. Data analysis was performed by Stata 11.0. Differences between HCV group and healthy control group in continuous and categorical variables were examined using conditioned logistic regression. Subgroups of non- and low-responders versus normal- and high-responders were evaluated in relation to demography characteristics, biochemical indicators, liver disease statues and HCV RNA. A Student's t test or one-way ANOVA were used to compare the average anti-HBs titer between different subgroups. Fisher's exact test was used to compare the response rates. Nonparametric test was used to compare immunodotting spots. Sperman rank correlation analysis was used to evaluate the correlation between immunodotting spots and anti-HBs. For all these comparisons, a two-side P<0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for HCV group were as follows: (1) aged ≥ 22 years and Han nationality; (2) no history of hepatitis B vaccination; (3) not-in-treatment patients with anti-HCV and HCV RNA positive; (4) diagnosis of chronic hepatitis C on the basis of self-reported history of HCV infection (more than 6 months) and screening tests for inclusion; (5) negative for HBsAg, anti-HBs, hepatitis B e antigen (HBeAg), antibody to hepatitis B e antigen (anti-HBe) and antibody to hepatitis B core antigen (anti-HBc).

Inclusion criteria for healthy control group were as follows: (1) aged ≥ 22 years and Han nationality; (2) no history of hepatitis B vaccination; (3) negative for anti-HCV and HCV RNA; (4) negative for HBsAg, anti-HBs, HBeAg, anti-HBe and anti-HBc; (5) no self-reported acute and chronic diseases.

Exclusion Criteria:

* (1) allergy to any vaccine component; (2) pregnancy or lactation; (3) axillary temperature ≥38℃ in the past three days, acute disease in the past seven days or vaccination history of any vaccine in the past four weeks; (4) suffering from diseases that may influence immune function, such as severe cirrhosis with Child-Pugh score >5, renal failure, bleeding diathesis, malignant tumor and HIV infection; (5) have received or being taking antiviral treatment; (6) chronic liver diseases except causing by HCV.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Antibody to the hepatitis B surface antigen response and cytokine response to hepatitis B vaccination in patients with chronic HCV. | one month after the third dose of vaccination
  Three doses of hepatitis B vaccine made by Recombinant DNA Techniques in Saccharomyces Cerevisiae (20 μg HBsAg/1.0ml per dose, Shenzhen Kangtai Biological Products Co., Ltd., Shenzhen, Guangdong Province, China) were given intramuscularly in the deltoid region to all participants at 0, 1 and 6 months respectively. Blood samples from the participants were collected one month after the third dose of vaccination. Anti-HBs was assayed by Abbott Chemiluminesent Microparticle ImmunoAssay (CMIA) (Abbott Ireland Diagnostics Division, Sligo, Ireland) one month after the first and the third dose of vaccination. Spot-forming Cells (SFCs) were enumerated with ImmunoSpotTM system (Cellular Technology Ltd.). Differences between HCV group and healthy control group in anti-HBs and immunodotting spots were examined.

SECONDARY OUTCOMES:
The occurrence and severity of solicited local reactions at the injection site, solicited systemic reactions, and any unsolicited adverse after hepatitis B vaccination in patients with chronic HCV | from the first dose of vaccination to one month after the third dose of vaccination
  Participants were provided with diary cards to record the occurrence and severity of solicited local reactions at the injection site (pain, induration, erythema, edema, pruritus) during 7 days after vaccination, solicited systemic reactions (fever, headache, fatigued, cough, myalgia, asthenia, vertigo, diarrhea), and any unsolicited adverse during 29 days after vaccination.